CLINICAL TRIAL: NCT04938609
Title: Neoadjuvant Immunoradiotherapy in Head & Neck Cancer (NIRT 2-HNC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Providence Cancer Center, Earle A. Chiles Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020000720 NIRT 2
Record Dates: First submitted 2021-06-09; First posted 2021-06-24 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; radiation; surgery; pembrolizumab; Phase 2; immunotherapy; antibodies
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + SBRT + Surgery (Experimental): Pembrolizumab administration (3 dose) every 3 weeks and 1 dose before radiation (5 days) therapy followed by an additional administration of Pembrolizumab (2 doses) prior to restaging and surgical resection followed by risk-adapted adjuvant therapy, per standard of care. Patient will then be treated with adjuvant pembrolizumab every 3 weeks for 14 additional doses (17 doses total)
  Interventions: Drug: Pembrolizumab; Radiation: Stereotactic Body Radiation Therapy (5 days); Procedure: Surgical Resection

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a humanized anti-PD-1 mAb of the IgG4/kappa isotype with a stabilizing S228P sequence alteration in the Fc region.
  Other Names: Keytruda
Radiation: Stereotactic Body Radiation Therapy (5 days) — 8Gy x 3 (Mon-Fri) GTV+3mm
Procedure: Surgical Resection — Surgical Resection of Tumor

SUMMARY:
The purpose of this study is to evaluate the efficacy of neoadjuvant immunoradiotherapy (NIRT) prior to surgery for the treatment of stage III and IVA HPV- HNSCC.

DETAILED DESCRIPTION:
This clinical trial uses pembrolizumab and radiotherapy prior to definitive surgical resection of tumors in patients with Head and Neck Squamous Cell Carcinoma (OHNSCC) with the primary objective of determining the safety and efficacy of preoperative immunoradiotherapy. In addition, tumor tissue, microbiome samples, and peripheral blood will be obtained for exploratory immunologic end points including measurements of tumor infiltrating immune cell populations based on flow cytometry and immunohistochemistry as well as circulating immunological parameters.

Estimated duration of 52 weeks: neoadjuvant immunoradiotherapy +/- surgery at week 7, followed by risk adapted adjuvant therapy, per standard of care. Patients will then be treated with adjuvant pembrolizumab every 3 weeks for 14 additional doses (17 doses total).

Phase II efficacy study (n = 28, total) to assess rate of down-staging after neoadjuvant immunoradiotherapy using Simon's two-stage design (futility assessment at n = 12).

Phase I studied nivolumab in 10 patients with HPV+ HNSCC, the results of which suggest that the combination is safe and efficacious. The phase II portion of study will evaluate the efficacy of neoadjuvant pembrolizumab in combination with SBRT as a safe means to down-stage HNSCC prior to surgical resection, improve quality of life, and enhance local control and overall survival. Patients will be followed for disease free and overall survival at 5 years.

Eligible patients may be enrolled unless a rate of unplanned surgical delay attributed to immunoradiotherapy is found to exceed 33% after enrollment of the first 10 patients. We estimate at least 2 patients per month will be enrolled. Time to full accrual is estimated as 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent.
2. Histologically confirmed diagnosis of stage III-IVA HPV-negative HNSCC who are planned for surgical resection and in the opinion of the investigator are able to safely undergo neoadjuvant anti-PD-1 and radiation will be enrolled in this study. Oral cavity, hypopharynx, and larynx cancer are not required to undergo HPV testing by p16 IHC as by convention these tumor locations are assumed to be HPV-negative

   Male participants:
3. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 75 days, corresponding to time needed to eliminate any study treatment) plus an additional 120 days (a spermatogenesis cycle) after the last dose of study treatment and refrain from donating sperm during this period.

   Female participants:
4. A female participant is eligible to participate if she is not pregnant (see Appendix 3),or breastfeeding and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 75 days (corresponding to time needed to eliminate any study treatment) plus 30 days (a menstruation cycle) after the last dose of study treatment.
5. The participant must provide (or legally acceptable representative if applicable) written informed consent for the trial.
6. Have provided archival tumor tissue sample collected within the last 6 months or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

   Note: If submitting unstained slides, slides should be submitted to the testing laboratory within 14 days from the date slides are cut. For archival tissue samples collected >6 months from screening, PI approval is required.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 10 days prior to the date of enrollment
8. Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

1. A WOCBP who has a positive serum or urine pregnancy test within 72 hours prior to first dose of pembrolizumab (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to enrollment

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Has received prior radiotherapy to the head and neck region.
5. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) or other solid tumor or hematologic malignancy that have undergone potentially curative therapy outside of the head and neck are not excluded.
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV) testing is not required unless mandated by local health authority
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Has a known history of active TB (Bacillus Tuberculosis). testing is not required unless mandated by local health authority
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
20. Patients with T1,T2 and T3 larynx cancer are excluded.
21. Patients with prior history of solid organ and/or allo-transplantation.
22. Patients with pre-existing neuropathy of grade 2 or higher peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2027-01-11 (Estimated); Study Completion 2031-01-11 (Estimated)

PRIMARY OUTCOMES:
To determine the pathologic response rate (MPR + pCR) at time of surgery | 52 weeks
  Prior to surgery neoadjuvant immunoradiotherapy (NIRT) with stereotactic body radiation therapy (SBRT) + pembrolizumab in stage III-IVA HPV-negative HNSCC patients.

SECONDARY OUTCOMES:
Overall Response Rate | 5 years
  Number of patients who have a partial or complete response to treatment per RECIST 1.1.
Clinical swallowing evaluation assessed by VFSS | 5 years
  Clinical swallowing evaluation using the Video Fluoroscopic Swallowing Study (VFSS)
Quality of Life assessed by PSS-HN | 5 years
  Quality of life using the Performance Status Scale for Head and Neck Cancer (PSS-HN)
Quality of Life assessed by FACT-H&N | 5 years
  Quality of life using Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-H&N)
Quality of Life assessed by MDASI-HN | 5 years
  Quality of life using the MD Anderson Symptom Inventory for head and neck cancer (MDASI-HN) module.
Quality of Life assessed by Eat-10 | 5 year
  Quality of life using the Eating Assessment Tool (Eat-10)
Quality of Life assessed by FOIS | 5 years
  Quality of life using the Functional Oral Intake Scale FOIS
Quality of Life assessed by UW-QOL | 5 years
  Quality of life using the University of Washington Quality of Life Questionnaire (UW-QOL)
Adverse events | From time of informed consent through 90 days after the last study treatment
  Frequency, duration, and severity of adverse events
Surgical Complications | 30 days post-op
  Post surgery: Clavien-Dindo classification for grading surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: R. Bryan Bell, MD, DDS, FACS, Principal Investigator — Providence Health & Services
Locations (3):
- United States (3):
  - University of San Diego, San Diego, California
  - Portland Providence Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon